CLINICAL TRIAL: NCT05378009
Title: Functional Dyspepsia Response to Relaxation Therapy Alone or Combined With Physical Activity
Brief Title: Functional Dyspepsia Response to Relaxation Therapy and Physical Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003657
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): This FD women group will include 30 females who will be treated for 8 weeks with oral proton pump inhibitors (taken one time daily with 40 mg pantoprazole-tablet dose), Benson relaxation daily sessions (twenty minutes at morning time and another 20 minutes at the evening time), physical activity ( five session per the week conducted on treadmill, 30 minutes in the first treatment month and 40 minutes in the second treatment month)
  Interventions: Behavioral: relaxation and physical activity
- Group B (Active Comparator): This FD women group will include 30 females who will be treated for 8 weeks with oral proton pump inhibitors (taken one time daily with 40 mg pantoprazole-tablet dose) and Benson relaxation daily sessions (twenty minutes at morning time and another 20 minutes at the evening time)
  Interventions: Behavioral: relaxation

INTERVENTIONS:
Behavioral: relaxation and physical activity — This FD women group will include 30 females who will be treated for 8 weeks with oral proton pump inhibitors (taken one time daily with 40 mg pantoprazole-tablet dose), Benson relaxation daily sessions (twenty minutes at morning time and another 20 minutes at the evening time), physical activity ( five session per the week conducted on treadmill, 30 minutes in the first treatment month and 40 minutes in the second treatment month)
  Arms: group A
Behavioral: relaxation — This FD women group will include 30 females who will be treated for 8 weeks with oral proton pump inhibitors (taken one time daily with 40 mg pantoprazole-tablet dose) and Benson relaxation daily sessions (twenty minutes at morning time and another 20 minutes at the evening time)
  Arms: Group B

SUMMARY:
Functional dyspepsia (FD) is a common gastrointestinal disease with high morbidity. Due to the drop in estrogen level, perimenopausal women with FD (PMFD) have an increase in emotional disorders such as depression, anxiety and sleep disorder.

DETAILED DESCRIPTION:
the research will include 30 FD women during their perimenopause to receive for 8 weeks the following: relaxation therapy (Benson relaxation), physical exercise (on treadmill), and proton pump inhibitors. Also, the research will include another 30 FD women during their perimenopause to receive for 8 weeks the following: relaxation therapy (Benson relaxation) and proton pump inhibitors

ELIGIBILITY:
Inclusion Criteria:

* perimenopausal women With FD symptoms

Exclusion Criteria:

* other gastrointestinal disease
* Cardiovascular, metabolic, respiratory, renal complaints
* Pregnancy
* Women in Lactation
* neurological / Psychic Women

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
cortisol | It will be measured after 8 weeks
  stress hormone will be measured in serum

SECONDARY OUTCOMES:
Glasgow dyspepsia severity score | It will be measured after 8 weeks
  it is questionnaire assessing severity of dyspepsia
Visual analogue scale | It will be measured after 8 weeks
  it is a scale for assessment of severity of abdominal syymptoms
depression anxiety stress scales-42 | It will be measured after 8 weeks
  it is a 42 item self-report scale designed to measure the negative emotional states of depression, anxiety and stress
Pittsburgh sleep quality index | It will be measured after 8 weeks
  it is a questionnaire for sleep quality assessment
Estradiol | It will be measured after 8 weeks
  one of endogenous estrogen in the serum of women

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt